CLINICAL TRIAL: NCT00449488
Title: A Prospective, Randomised, Clinical Study to Examine the Effects of a Single Bolus Erythropoietin on Left Ventricular Function in Patients With an Acute Myocardial Infarction
Brief Title: Clinical Study to Examine the Effects of Erythropoietin on Left Ventricular Function After Acute Myocardial Infarction
Acronym: HEBEIII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: The Interuniversity Cardiology Institute of the Netherlands (Other Government); Janssen-Cilag Ltd. (Industry)
Responsible Party: A.A. Voors, University Medical Center Groningen, department of Cardiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B213; ISRCTN46528154
Record Dates: First submitted 2007-03-18; First posted 2007-03-20 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Myocardial Infarction
Keywords: erythropoietin; myocardial infarction; PCI; left ventricular function
MeSH Terms: conditions — Myocardial Infarction | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention)
- Epoetin alfa (Active Comparator): i.v bolus 60.000 IU epoetin alfa
  Interventions: Drug: epoetin alfa

INTERVENTIONS:
Drug: epoetin alfa — epoetin alfa 60.000 IU one i.v. bolus
  Other Names: Eprex
  Arms: Epoetin alfa

SUMMARY:
The primary objective of this study is to establish the effects of a single bolus of EPO, administered within three hours after a primary PCI for a first acute myocardial infarction, on left ventricular function.

DETAILED DESCRIPTION:
Erythropoetin (EPO) is commonly known as an effective treatment for anemia. However, several important extra-hematopoeitic effects of EPO are suggested which might be beneficial in the setting of an acute myocardial infarction, such as a reduction of apoptosis and stimulation of neovascularisation. Recent animal studies provided very consistent evidence for a reduced infarct size and improved left ventricular function caused by EPO administration. However, clinical studies with EPO in non-anemic patients are scarce.

We performed a safety study in our department on the effects of a single bolus of EPO in patients with an acute myocardial infarction. Serum EPO levels increased a 200-fold and EPO administration was not associated with hypertension, nor with an increase in thrombocytes or thrombotic events.

In conclusion, experimental data clearly showed that a single bolus of EPO after the onset of an acute myocardial infarction reduced myocardial infarct size, and improved left ventricular function. In our safety study, EPO administration in patients with an acute myocardial infarction was safe and well tolerated.

This will be a PROBE (Prospective, Randomised, Open label study with Blinded Endpoint) designed study, in wich one group will receive one bolus of EPO 60.000 IU) intravenously within 3 hours after the primary PCI procedure and the other group will receive standard therapy. After 6 weeks left ventricular ejection fraction will be evaluated by planar radionuclide ventriculography.

ELIGIBILITY:
Inclusion Criteria:

Successful primary PCI (TIMI 2/3) for a first acute myocardial infarction, diagnosed by:

* chest pain suggestive for acute myocardial infarction
* symptom onset < 12 hour before hospital admission, or < 24 hour in case ongoing ischemia
* ECG with ST-T segment elevation > 1 mV in 2 or more leads
* TIMI flow 0/1 before primary PCI on diagnostic coronary angiography;

Exclusion Criteria:

* Hemoglobin levels > 10.6 mmol/L;
* Anticipated additional revascularisation within 4 months;
* Cardiogenic shock;
* Presence of other serious medical conditions
* Pregnancy/breast feeding
* Malignant hypertension
* End stage renal failure (creatinin > 220 micromol/l)
* Previous treatment with rh-EPO
* Blood transfusion <12 weeks prior to randomisation
* Polycythemia vera
* Previous acute myocardial infarction
* Concomitant inflammatory or malignant disease
* Recent trauma or major surgery
* Unwilling to sign informed consent
* Atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2007-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction 6 weeks after primary PCI, measured with planar radionuclide ventriculography | 6 weeks

SECONDARY OUTCOMES:
Safety, myocardial infarct size, and cardiovascular events at 6 weeks after a single bolus of EPO | Cardiovascular Events

CONTACTS AND LOCATIONS:
Overall Officials: A A Voors, MD,PhD, Principal Investigator — University Medical Center Groningen; F Zijlstra, MD,PhD,FACC, Principal Investigator — University Medical Center Groningen; DJ van Veldhuisen, MD,PhD,FACC, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Background] Belonje AM, Voors AA, van Gilst WH, Anker SD, Slart RH, Tio RA, Zijlstra F, van Veldhuisen DJ; HEBE III investigators. Effects of erythropoietin after an acute myocardial infarction: rationale and study design of a prospective, randomized, clinical trial (HEBE III). Am Heart J. 2008 May;155(5):817-22. doi: 10.1016/j.ahj.2007.12.036. PMID 18440327
- [Derived] Voors AA, Belonje AM, Zijlstra F, Hillege HL, Anker SD, Slart RH, Tio RA, van 't Hof A, Jukema JW, Peels HO, Henriques JP, Ten Berg JM, Vos J, van Gilst WH, van Veldhuisen DJ; HEBE III Investigators. A single dose of erythropoietin in ST-elevation myocardial infarction. Eur Heart J. 2010 Nov;31(21):2593-600. doi: 10.1093/eurheartj/ehq304. Epub 2010 Aug 29. PMID 20802250